CLINICAL TRIAL: NCT01067079
Title: A Phase III, Single Center, Open Label, Follow-up Immunogenicity Study in Subjects Who Previously Received Post-exposure Rabies Vaccine According to the Essen or 2:1:1 (Zagreb) Schedule
Brief Title: Single Center, Open Label, Follow up Study in Subjects Who Previously Received Rabies Vaccine as Simulated Post-Exposure Regimen
Status: Terminated | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: M49P8E1
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Rabies
Keywords: Rabies vaccine; Long-term Immunogenicity
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Arm 1
  Interventions: Other: No vaccine administered; subjects only have blood sampling for immunogenicity

INTERVENTIONS:
Other: No vaccine administered; subjects only have blood sampling for immunogenicity — No vaccine administered; subjects only have blood sampling for

SUMMARY:
This study will evaluate the immunogenicity of rabies vaccine at 13 months, 3 year and 5 years after initial vaccination, administered in two different post-exposure vaccination schedules

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects who received complete vaccine series in accordance to the designated vaccination schedule in the previous M49P8 study

Exclusion Criteria:

* Any disease condition, that in the opinion of investigator may interfere with subjects ability to participate in the study.
* Receipt of additional doses of rabies vaccine after completion of initial vaccine series.
* For additional entry criteria please refer to protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who received complete vaccine series in accordance to the designated vaccination schedule in the previous M49P8 study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Rabies virus neutralizing antibody(RVNA) responses 13months, 3 years and 5 years after completion of initial vaccination series as evaluated by percentage of subjects with RVNA greater than or equal to 0.5 IU/mL | 13 months, 3 years and 5 years after initial vaccination

SECONDARY OUTCOMES:
Rabies virus neutralizing antibody(RVNA) responses 13months, 3 years and 5 years after completion of initial vaccination series as evaluated by geometric mean concentration | 13months, 3 years and 5years after initial vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jizhou County, Hebei, China

REFERENCES:
- [Derived] Ma J, Wang H, Li J, Chang L, Xie Y, Liu Z, Zhao Y, Malerczyk C. A randomized open-labeled study to demonstrate the non-inferiority of purified chick-embryo cell rabies vaccine administered in the Zagreb regimen (2-1-1) compared with the Essen regimen in Chinese adults. Hum Vaccin Immunother. 2014;10(10):2805-12. doi: 10.4161/21645515.2014.972773. PMID 25483635